CLINICAL TRIAL: NCT04462471
Title: A Phase Ib Trial of Vemurafenib Plus Copanlisib to Enhance Radioiodine Avidity in Radioiodine-Refractory Thyroid Cancers
Brief Title: Vemurafenib Plus Copanlisib in Radioiodine-Refractory (RAIR) Thyroid Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-053
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Carcinoma; Thyroid Cancer; Thyroid Cancer, Follicular; Thyroid Cancer (Follicular Cell); Thyroid Cancer, Papillary; BRAF V600E Mutation Positive
Keywords: thyroid carcinoma of follicular origin; thyroid cancer; thyroid cancer, follicular; thyroid cancer, papillary; thyroid cancer, poorly differentiated; BRAF V600; RAIR disease; Memorial Sloan Kettering Cancer Center; 20-053
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid cancer, follicular; Thyroid Cancer, Papillary | interventions — Vemurafenib; copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with thyroid cancer (Experimental): Eligible participants will have a diagnosis of BRAF mutant RAIR thyroid cancer
  Interventions: Diagnostic Test: I-124 PET/CT lesion dosimetry; Drug: Vemurafenib; Drug: Copanlisib

INTERVENTIONS:
Diagnostic Test: I-124 PET/CT lesion dosimetry — I-124 PET/CT scans will be performed during this process to quantify baseline RAI avidity in index metastatic lesion(s)
Drug: Vemurafenib — Dose level 1 & 2: 960 mg PO bid Dose level -1: 720 mg PO bid Dose level -2: 480 mg PO bid
Drug: Copanlisib — Dose level 2: 60 mg IV weekly Dose level 1, -1, -2: 45 mg IV weekly

SUMMARY:
The purpose of this study is to develop a new drug treatment to reverse tumor resistance to radioiodine in BRAF mutant tumors so that radioiodine can be given to shrink tumors. This study is also being done to find out the highest doses of copanlisib and vemurafenib that, when given in combination, do not cause serious side effects, and whether the study treatment will make radioiodine therapy work better in patients with BRAF-mutant thyroid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed thyroid carcinoma of follicular origin (including papillary, follicular, and poorly differentiated subtypes and their respective variants).
* A tumor sample (primary, recurrent, or metastatic tumors) possessing a BRAF V600 mutation, as confirmed in a CLIA-certified laboratory or using an FDA-approved assay
* Measurable disease by RECIST v1.1 (tumors in previously irradiated fields may be considered measurable if there is evidence of tumor progression after radiation treatment)
* RAIR disease, as defined by any one of the following:

  * A metastatic lesion that is not RAI-avid on a diagnostic radioiodine scan
  * An RAI-avid lesion that remained stable in size or progressed despite RAI treatment before entry in this study (there are no size limitations for the index lesion used to satisfy this entry criterion)
  * The presence of at least 1 FDG-avid lesion
* No receipt of treatment for thyroid cancer, defined as:

  * No I-131 therapy < 6 months before initiation of the protocol (time of initiation of the protocol is defined as the first day of drug therapy with vemurafenib and copanlisib); diagnostic activities of I-131 (0-10m Ci) are allowed within 6months of initiating the protocol
  * No external beam radiation therapy <4 weeks before initiation of the protocol
  * No chemotherapy or targeted therapy including TKIs <4 weeks (or <5 half lives of the drug) before the initiation of this protocol
* Age of ≥ 18 years
* ECOG performance status ≤ 2 or Karnofsky Performance Score (KPS) ≥ 70%
* Tissue from the primary tumor or metastases available for correlative studies. Either a paraffin block or at least 20 unstained slides are acceptable (30 unstained slides is ideal); if <20 unstained slides are available, and a paraffin block is not available, the patient may be able to participate at the discretion of the investigator
* Able to swallow and retain an orally administered pill without any clinically significant gastrointestinal abnormalities that may alter absorption, such as malabsorption syndrome or major resection of the stomach or bowels
* Agree to undergo 2 research biopsies of (a) malignant lesion(s). Tumor tissue obtained before study consent or treatment can also be submitted in lieu of performance of the first pretreatment biopsy if the Principal Investigator deems it to be of sufficient quantity/quality/timeliness (tumor tissue obtained more than 3 years from time of study consent would not be eligible). Patients may be exempt from biopsy if (1) the investigator or person performing the biopsy judges that no tumor is accessible for biopsy, (2) the investigator or person performing the biopsy feels that the biopsy poses too great of a risk to the patient, or (3) the patient's platelet count is <100,000/mcL or the patient cannot be safely removed from anticoagulation therapy (if the anticoagulation therapy needs to be temporarily held for the biopsy procedure). If the investigator deems a second research biopsy to be high risk, the patient may be exempt from the second biopsy.
* Screening laboratory values meeting the following criteria:

  * WBC ≥ 2000/µL
  * Neutrophils ≥ 1500/µL
  * Platelets ≥ 100 × 10^3/µL
  * Hemoglobin >9.0 g/dL
  * Lipase ≤ 1.5 × ULN
  * AST/ALT ≤ 3 × ULN
  * Total bilirubin ≤ 1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin <3.0 mg/dL)
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

Female CrCl = (140 - age in years) x weight in kg x 0.85 / 82 x serum creatinine in mg/dL

Male CrCl = (140 - age in years) x weight in kg x 1.00 / 72 x serum creatinine in mg/dL

Exclusion Criteria:

* Untreated metastatic brain or leptomeningeal tumors (metastatic brain or leptomeningeal tumors treated with radiation and/or surgery are allowed)
* Prior malignancy if diagnosed and treated within 2 years of trial drug initiation (with the exception of nonmelanoma skin cancers or Stage I cancers treated with curative intent).Patients may be included if they have completed therapy for a prior malignancy >2 years before drug initiation and currently have no evidence of disease
* Inability to follow a low-iodine diet or requiring a medication with a high content of iodide (amiodarone)
* Current congestive heart failure class >2, as defined by the New York Heart Association functional classification system
* Myocardial infarction < 6 months before the initiation of protocol
* Unstable angina (angina symptoms at rest) or new-onset angina (begun within the last 3 months)
* Uncontrolled hypertension (blood pressure >150/90, despite optimal medical management)
* Uncontrolled type I or II diabetes mellitus, as judged by the investigator, or Hgb A1C of >8.5
* Arterial or venous thrombotic event or embolic event, such as a cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism, within 3 months before the start of study medication
* Nonhealing wound, ulcer, or bone fracture (tumor-related nonhealing wounds are allowed)
* Active, clinically serious infections CTCAE v5.0 grade >2
* History of concurrent condition of interstitial lung disease and/or severely impaired lung function
* Known history of HIV infection (all patients must be screened for HIV up to 28 days before start of study)
* Seizure disorder requiring medication
* Therapy with a prohibited concomitant medication that cannot be temporarily held (at least 2 weeks before initiation of vemurafenib plus copanlisib until 1 week after the last dose) or replaced with a nonprohibited concomitant medication
* Systemic corticosteroid therapy at a daily dose >15 mg prednisone or equivalent (previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days before study registration)
* Cytomegalovirus (CMV) PCR-positive at baseline
* Evidence or history of a bleeding diathesis or any hemorrhage or bleeding CTCAE v5.0 grade ≥ 3 within 4 weeks before the start of study protocol
* HBV or HCV infection. All patients must be screened for HBV and HCV up to 28 days before the start of study medication using the routine hepatitis virus laboratorial panel. Patients positive for HBsAg or HBcAb will be eligible if they are negative for HBV-DNA (these patients should receive prophylactic HBV antiviral therapy). Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA
* Known hypersensitivity to any of the test drugs, test drug classes, or excipients in the formulation
* Substance abuse or medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Patients who are pregnant
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 6 months after the last administration of study treatment. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment. In cases of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone-level assessment (FSH level in the postmenopausal range) is this acceptable
  * Male sterilization (at least 6 months before screening). The vasectomized male partner should be the sole partner for that patient
  * Use of oral, injected, or implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system or other forms of hormonal contraception that have comparable efficacy (failure rate <1%)-for example, hormone vaginal ring or transdermal hormone contraception. Note: In cases of use of oral contraception, women should have been stable, on the same pill for a minimum of 3 months before taking study treatment
  * Women are considered postmenopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks ago. In cases of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone-level assessment is she considered not of child-bearing potential.
* Sexually active men, unless they use a condom during intercourse while on treatment and for 6 months after stopping treatment with study drugs (men should not father a child in this period). A condom is required to be used by vasectomized men as well during intercourse to prevent delivery of the drug via semen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan L Ho, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan-Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Mauguen A, Grewal RK, Augensen F, Abusamra M, Mahajan S, Jayaprakasam VS, Osborne J, Haque S, Wong BZY, Ghossein RA, Fagin J, Schӧder H, Tuttle RM, Ho A, Humm JL, Larson SM. The use of single-timepoint images to link administered radioiodine activity (MBq) to a prescribed lesion radiation-absorbed dose (cGy): a regression-based prediction interval tool for the management of well-differentiated thyroid cancer patients. Eur J Nucl Med Mol Imaging. 2023 Aug;50(10):2971-2983. doi: 10.1007/s00259-023-06240-1. Epub 2023 May 12. PMID 37171634
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Dose Level 1: Vemurafenib 960mg, Copanlisib 45mg
- Dose Level 2: Dose Level 2: Vemurafenib 960mg, Copanlisib 60mg
- Dose Level -1: Dose Level -1: Vemurafenib 720mg, Copanlisib 45mg
- Dose Level -2: Dose Level -2: Vemurafenib 480mg, Copanlisib 45mg
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -1 | Dose Level -2
Started | 4 | 4 | 0 | 0
Completed | 3 | 3 | 0 | 0
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Disease progression | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were treated on Dose Level -1 and Dose Level -2
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -1 | Dose Level -2 | Total
Number analyzed (Participants) | 4 | 4 | 0 | 0 | 8
Age, Continuous [Mean (Full Range); unit: years] | 56 [44 to 66] | 54 [42 to 73] |  |  | 55 [42 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 |  |  | 2
  Male | 3 | 3 |  |  | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 |  |  | 1
  Not Hispanic or Latino | 4 | 3 |  |  | 7
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 |  |  | 0
  White | 4 | 4 |  |  | 8
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 |  |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: The primary objective of this study is to determine the MTD of vemurafenib plus copanlisib inpatients with advanced BRAF mutant RAIR thyroid cancer. The MTD is defined as the highest dose at which no more than 1 of 6 patients treated at that dose experience a DLT.
Time Frame: 6 months
Population: Study closed to low accrual
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -1 | Dose Level -2
Number analyzed (Participants) | 4 | 4 | 0 | 0
Participants
  Experienced DLT | 0 | 0 | 0 | 0
  Did not experience DLT | 4 | 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Participants were not treated on Dose Level -1 or Dose Level -2
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level -1 | Dose Level -2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/4 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=4) | Dose Level -1 (N=0) | Dose Level -2 (N=0)
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | NA | NA
Anemia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Creatinine increased (Investigations) | 0 | 1 | NA | NA
Fever (General disorders) | 0 | 1 | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 1 | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 1 | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=4) | Dose Level -1 (N=0) | Dose Level -2 (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 0 | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | NA | NA
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 0 | NA | NA
Blood bilirubin increased (Investigations) | 0 | 1 | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | NA | NA
Creatinine increased (Investigations) | 1 | 3 | NA | NA
Diarrhea (Gastrointestinal disorders) | 2 | 1 | NA | NA
Dry mouth (Gastrointestinal disorders) | 1 | 0 | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Dysgeusia (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Fatigue (General disorders) | 1 | 2 | NA | NA
Fever (General disorders) | 1 | 0 | NA | NA
Headache (Nervous system disorders) | 1 | 1 | NA | NA
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | NA | NA
Hypertension (Metabolism and nutrition disorders) | 1 | 1 | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Hypothyroidism (Endocrine disorders) | 1 | 0 | NA | NA
Lipase increased (Investigations) | 1 | 0 | NA | NA
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Nausea (Gastrointestinal disorders) | 1 | 1 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA | NA
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA
Palpitations (Cardiac disorders) | 1 | 0 | NA | NA
Photophobia (Eye disorders) | 0 | 1 | NA | NA
Platelet count decreased (Investigations) | 0 | 1 | NA | NA
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | NA | NA
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 1 | NA | NA
Urinary frequency (Renal and urinary disorders) | 1 | 0 | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 1 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT04462471/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT04462471/ICF_001.pdf